CLINICAL TRIAL: NCT02731768
Title: Using Technology to Enhance Social Support for Weight Loss in Adults: The NETworks (Nutrition, Exercise, and Technology) Pilot Randomized Controlled Trial
Brief Title: Nutrition, Exercise, and Technology for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1205
Record Dates: First submitted 2016-02-23; First posted 2016-04-08 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Participants will receive an evidence-based behavioral weight control program focused on physical activity and reducing caloric intake. They will be provided with a Fitbit Zip and digital body weight scale for self-monitoring of physical activity and body weight, respectively. They will track caloric intake via the MyFitnessPal smartphone application. They will have access to a study website and attend weekly, in-person group counseling sessions.
  Interventions: Behavioral: Standard; Device: Fitbit Zip; Device: Digital body weight scale
- Social support-enhanced (Experimental): Participants will receive the same intervention components as the Standard group, as well as two extra Fitbit Zips and digital body weight scales to share with up to two persons in their social circle who will be invited to serve as their support partners.
  Interventions: Behavioral: Social support-enhanced; Device: Fitbit Zip; Device: Digital body weight scale

INTERVENTIONS:
Behavioral: Standard — Participants will receive an evidence-based behavioral weight control program focused on physical activity and reducing caloric intake. They will be provided with a Fitbit Zip and digital body weight scale for self-monitoring of physical activity and body weight, respectively.They will track caloric intake via the MyFitnessPal smartphone application. They will have access to a study website and attend weekly, in-person group counseling sessions.
  Arms: Standard
Behavioral: Social support-enhanced — Participants will receive the same intervention components as the Standard group.Participants will also be provided with two extra Fitbit Zips and digital body weight scales to share with up to two persons in their social circle who will be invited to serve as their support partners.
  Arms: Social support-enhanced
Device: Fitbit Zip
Device: Digital body weight scale

SUMMARY:
The purpose of this study is to evaluate whether a social support-enhanced, technology-based, behavioral weight control intervention can improve weight loss over existing best practices.

DETAILED DESCRIPTION:
This 4-month randomized controlled trial is designed to investigate the short-term efficacy and feasibility of a novel, social support-enhanced behavioral weight control intervention. Participants will be recruited via email listservs, fliers, and word of mouth. They will be randomized to a standard behavioral weight control treatment (SBT) or a social support-enhanced behavioral weight control treatment which receives the same intervention as SBT plus social support resources (specifically, additional self-monitoring technologies) for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 kg/m2 and 55 kg/m2
* Age 18 years or older
* Access to a computer with an Internet connection
* Smartphone ownership (Android or iOS)
* Willing to be randomized to either one of the two study groups
* Only one member of the same household eligible to participate

Exclusion Criteria:

* Currently lactating, pregnant, or planning to become pregnant during the length of the study
* Been diagnosed with type 1 or type 2 diabetes
* Medical or physical contraindications or limitations for engaging in physical activity
* History of major medical or psychiatric conditions
* Recent changes in medication known to affect weight
* Schedule that would prohibit or restrict attendance at a designated time for weekly in- person group meetings
* Currently participating in a weight management program
* Currently on medication that might affect weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Body Weight at 4 and 12 months | 0, 4, and 12 months

SECONDARY OUTCOMES:
Change from Baseline in Social Support for Exercise (Social Support for Exercise Scale) at 4 and 12 months | 0, 4, and 12 months
  Item scores will be averaged for each respective scale, yielding a final score for each participant. Change in average scores on each scale for each group will be computed.
Change from 2-month Autonomy Support (Important Other Climate Questionnaire) at 4 and 12 months | 2, 4, and 12 months
  Item scores will be averaged for the questionnaire, yielding a final score for each participant. Change in average scores for each group will be computed.
Change from Baseline Motivation for Weight Control (Treatment Self-regulation Questionnaire) at 4 months | 0 and 4 months
  Item scores will be averaged for the questionnaire on three subscales (autonomous, controlled, and amotivation), yielding a final score for each subscale for each participant. Change in average scores on each subscale for each group will be computed.
Change from Baseline Appropriate and Inappropriate Weight Control Practices (Weight Control Practices Checklist) at 4 and 12 months | 0, 4, and 12 months
  Total number of reported appropriate and inappropriate weight control practices will be computed for each participant. Change in the mean number of reported appropriate and inappropriate weight control practices for each group will be computed.
Change from Baseline Social Support Through Technology (2-item questionnaire - level of support and type of support through technology) at 4 and 12 months | 0, 4, and 12 months
  Change in average score on level of support obtained through technology for each group will be computed. Change in the type of support obtained through technology will be described using frequency counts and percentages for each group.
Change from Baseline Average Daily Step Counts measured via BodyMedia SenseWear armband (one-week time period) at 4 and 12 months | 0, 4, and 12 months
Change from Baseline in Social Support for Eating Habits (Social Support for Eating Habits Scale) at 4 and 12 months | 0, 4, and 12 months
Change from Baseline in Social Support for Weight Loss (Social Support for Weight Loss Scale) at 4 and 12 months | 0, 4, and 12 months

OTHER OUTCOMES:
Participant Satisfaction (Satisfaction Questionnaire) | 4 and 12 months
Participant Engagement-chat sessions | 0-4 months (all weeks)
  Number of chat sessions attended - recorded by investigator; number of days self-monitored diet on MyFitnessPal and physical activity on Fitbit - recorded by investigator; number of days self-monitored weight - self-reported via a weekly question on study website; number of log-ins to study website - objectively tracked via computer
Participant Engagement-diet and physical activity | 0-4 months (all weeks)
  Number of days self-monitored diet on MyFitnessPal and physical activity on Fitbit-recorded by investigator
Participant Engagement-weight | 0-4 months (all weeks)
  Number of days self-monitored weight-self-reported via a weekly question on study website
Participant Engagement-log-ins | 0-4 months (all weeks)
  Number of log-ins to study website-objectively tracked via computer

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Monroe, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be reported in aggregate.